CLINICAL TRIAL: NCT04028180
Title: Comparison Trial Between Two Repellent Products and a Positive Control Against Culicoides Nubeculosus Midges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCTEC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 928
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Midge Bites
MeSH Terms: interventions — Myelin Proteolipid Protein; picaridin

STUDY DESIGN:
Intervention Model Description: This was a single-centre, single-arm study with all participants testing one or more products at one dose. The control for each test was an untreated arm. There was no blinding or randomisation employed, since the outcome measures were based on midge behaviour. Repellent product testing took place in a laboratory setting using 15 participants, with a minimum of 3 of either gender per repellent product. Each participant tested at least one single product at one dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Midge Repellency (Experimental): Treatment of forearm with insect repellent and exposure to midges every 1 hour for 12 hours
  Interventions: Other: p-Menthane,3-8-diol (PMD) Topical Repellent; Other: Picaridin Topical Repellent

INTERVENTIONS:
Other: p-Menthane,3-8-diol (PMD) Topical Repellent — p-Menthane,3-8-diol (PMD) is a recommended active ingredient, which has been evaluated for safe use by the U.S. Environmental Protection Agency (USEPA)1. According to the USEPA laboratory exposure of animals to the active ingredient, PMD, this resulted in no adverse effects except eye irritation. The eye irritation potential of the finished product formulation has not been studied; therefore as a precaution, the products will be handled in the same way as the active ingredient. The researcher and participant must wear eye protection during application of the product and the potential for eye irritation is described in the Participant Information Sheet. . Participants will be excluded if they have a known allergy to any of the product ingredients, or any skin condition, which may affect their reaction to the product.
  There isn't a relevant intervention type hence why other is specified. It is to deter mosquitoes landing on the skin of a human.
  Other Names: NEO-PART PMD-XLTM (40% PMD) or NEO-PART PMD-XLTM (35% PMD)
Other: Picaridin Topical Repellent — Icaridin (trade names include Picaridin) is a known mosquito and midge repellent active ingredient. The active ingredient, Picaridin, has been classified as potentially mildly irritating/uncomfortable to the eyes - participants and researcher will wear safety glasses during handling of the products and the participants will be warned about the potential for irritation during the Informed Consent Procedure. Participants will also be excluded if they have a known allergy to any of the product ingredients, or any skin condition which may affect their reaction to the product.
  There isn't a relevant intervention type hence why other is specified. It is to deter mosquitoes landing on the skin of a human.
  Other Names: Smidge (20% Picaridin)

SUMMARY:
Comparison trial between two repellent products and a positive control against Culicoides nubeculosus midges. A single-centre laboratory setting study using healthy volunteers to test two insect repellent products and a positive control product against Culicoides nubeculosus midges. The test products are designed for use by the general public in areas where midge biting is likely.

DETAILED DESCRIPTION:
Mosquitoes, midges and other biting insects are vectors of extremely important diseases such as malaria, yellow fever, filariasis and many viruses and also may be of great nuisance value. The use of repellent products can provide added personal protection from disease transmission and nuisance bites. New effective repellents would offer an additional option for protection against biting insects. The aim of this study is to determine the effectiveness of two topically applied insect repellent products provided and one positive control against Culicoides nubeculosus. Culicoides nubeculosus is a common species of biting midges belonging to the family Ceratopogonidae. Culicoides midges are small biting flies found throughout the world, breeding primarily in moist, damp, muddy habitats. To develop their eggs, female Culicoides require a blood meal from warm-blooded vertebrates, most often a domesticated animal and humans. Culicoides are implicated in the transmission of multiple zoonotic diseases, such as bluetongue virus, African horse sickness, and bovine ephemeral fever, and their bites can be painful and can cause uncomfortable irritation to both humans and livestock.

This is a single-centre, single-arm study with all participants testing two formulations containing PMD and a positive control product containing Picaridin. The control for each test is an untreated arm. There is no blinding or randomisation employed, since the outcome measures are based on midge behaviour. Repellent product testing takes place in a laboratory setting using 7 participants (preferably gender balanced). Each participant will test both PMD formulations and a positive control product.

Volunteers will be consented prior to any screening procedures being undertaken. Volunteers who do not meet the criteria for eligibility will be excluded. In order to assess sensitivity in those volunteers who claim not to be sensitive to insect bites, volunteers will be given a bite test using the midge species used for testing. Participants can stop at any time without giving a reason for withdrawing. Data collected to the point of withdrawal will be used in the analysis of the study, unless the participant requests that their data is not used, in which case it will be removed from the database. Participants may also be removed at the discretion of the Chief Investigator, where continued participation may affect the safety of the participant or where there is a development of any condition which might interfere with study participation.

All adverse events and serious adverse events should be reported. Any questions concerning adverse event reporting should be directed to the chief investigator in the first instance.

The midges will be obtained from insecticide-susceptible reference strains held at the Pirbright Institute (Institute for Animal Health). They will be maintained at 22-24°C, 80-90% relative humidity, with a 12:12 hour photoperiod. Female midges will be host-seeking, of uniform age and 3-8 days post-emergence. Active host-seeking females will be selected to ensure a good response from the test midges using an aspirator or an appropriate airflow apparatus. Before the start of each test, the participant will insert a bare (control) left arm into the cage for 1 minute to assess biting activity of the midges. Only cages with at least 10 midges landing within one minute will be used in the tests. This same procedure is used to assess whether volunteers are attractive to the midges. The number of midges probing or biting the arm after 1 minute will be counted and recorded (to provide biting rate data of the control test for the Protective Efficacy endpoint) and the arm removed from the cage. Immediately after, the right (treated) arm is inserted into the cage for 1 minute. The number of midges probing or biting the arm after 1 minute will be counted and recorded. A further hour post-application of the repellent product, the left arm (control) of the volunteer is again inserted into the cage. The number of midges probing or biting the arm after 1 minute will be counted and recorded and the arm removed from the cage. If less than 10 midges land on the untreated arm during this 1 minute test the cage will be refreshed with new midges and the test repeated. Immediately after, the right (treated) arm is again inserted into the cage for 1 minute. The number of midges probing or biting the arm after 1 minute will be counted and recorded. This procedure will be repeated at hourly intervals throughout the test.

The products will be applied to the forearm between the wrist and elbow. Volunteers' forearm surface area is estimated using the WHO protocol for testing skin repellents below:

Area=1⁄(2 ) (C_W+C_E ) X D_EW

Where CW is the circumference of the wrist; CE is the circumference of the elbow; and DEW is the distance between the wrist and elbow in centimetres (cm). The dose is expressed using µl/cm2. The appropriate dose is then measured using a micropipette or balance and applied to the arm using a gloved finger.

Participants will be followed up within 72 hours after the test to assess any possible side effects or reactions to the bites and/or products.

With the exception of the Volunteer Questionnaire, which is completed by the participant, all data collected will be recorded in the case report forms (CRF) and signed by the person completing the CRF. The CRF is considered to be source data. Data to be collected are: Participant number and date of visit on every page, confirmation of informed consent, date of birth, eligibility details, bite test details (midge species, timing, 10 min and 72 h assessments), test visits (eligibility checklist, forearm measurement, product details, product application details, arm-in-cage testing data (time, fitness check, No. midges probing control arm, No. midges probing treated arm)) and adverse event monitoring. Data will be double entered and verified to ensure accuracy. CRFs will be kept in locked storage. Information in the database for each test will be linked to a relevant SOP, risk assessment, contract, and files of statistical analysis and location of report copy.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give fully informed consent;
* Able to understand and comply with the study procedures;
* Consider themselves to be in good general health;
* Male or female;
* Aged 18 to 65 years;
* Non-smokers or willing to refrain for 12 hours prior to and during each test;
* Willing to undergo a bite test with Culicoides nubeculosus midges with up to 72 hour follow-up.

Exclusion Criteria:

* Suspected or known to be sensitive or allergic to midge bites;
* Participated in an interventional study (other than a biting insect challenge study) in the previous 3 months;
* Participated in a biting insect challenge study in the previous 72 hours;
* Aware of having any cardiovascular or respiratory disorder (whether active or inactive) (e.g. asthma);
* Individuals with localized skin disorders affecting the forearm;
* Allergic to any of the test product ingredients;
* Extensive tattooing or other conditions of the forearm which would make interpretation of the bite test results difficult;
* Women who are pregnant, nursing or intending to become pregnant;
* Previous anaphylaxis;
* Aware of having a compromised immune system;(an immune system that is temporarily or permanently incapable of working at full capacity);
* Phobia of flying insects;
* Travelled to a mosquito-borne disease endemic area in the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Median Complete Protection Time | 12 hours
  The time between application of the repellent product and the occurrence of the first probe or bite in a 1 minute test, followed by a confirmatory probe or bite within 30 minutes.

SECONDARY OUTCOMES:
Protective Efficacy | 12 hours
  Protective Efficacy is expressed as the percentage of midges probing or biting at hourly intervals from the time of the repellent application to the end of the test.

CONTACTS AND LOCATIONS:
Overall Officials: James Logan, PhD, Study Chair — ARCTEC
Locations (1):
- Arctec at London School of Hygiene & Tropical Medicine, London, United Kingdom

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT04028180/Prot_SAP_000.pdf